CLINICAL TRIAL: NCT04400916
Title: Topical Use of Tranexamic Acid for Prevention of Subconjunctival Hemorrhage After Intravitreal Injections
Brief Title: Topical Tranexamic Acid After Intravitreal Injections
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Shiri Soudry MD, Attending faculty and vitreoretinal surgeon, Department of Ophthalmology, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0424-19-RMB
Record Dates: First submitted 2020-05-20; First posted 2020-05-26 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Subconjunctival Hemorrhage
MeSH Terms: interventions — Tranexamic Acid; Hanks Balanced Salt Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical tranexamic acid (Experimental)
  Interventions: Drug: Tranexamic acid
- Topical BSS (Placebo Comparator)
  Interventions: Other: Balanced Salt Solution

INTERVENTIONS:
Drug: Tranexamic acid — A single drop administered topically
  Arms: Topical tranexamic acid
Other: Balanced Salt Solution — A single drop administered topically
  Arms: Topical BSS

SUMMARY:
We aim to investigate whether topical administration of Tranexamic acid can reduce the occurence of subconjunctival hemorrahge after routine intravitreal injections for retinal conditions.

ELIGIBILITY:
Inclusion Criteria:

Subjects receiving intravitreal injections as part of their routine ophthalmological care

Exclusion Criteria:

Pregnancy, Oral contraceptives/HRT use, Known systemic autoimmune disease, Renal failure, active/suspected infection or inflammation in the treated eye, subconjunctival hemorrahge prior to inclusion, History of subarachnoid hemorrahge, thromboembolic events, increased risk for thromboembolic events, known sensitivity to the study drug

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Subconjunctival hemorrahge | 3 days

IPD SHARING:
Plan to Share IPD: No